CLINICAL TRIAL: NCT02799628
Title: Positive Appraisal Improve Trust Between Patients and Therapists, and Change Treatment Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TYGH104046
Record Dates: First submitted 2016-06-05; First posted 2016-06-15 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Trust; Low Back Pain
Keywords: Trust; Low Back Pain; Treatment Outcome
MeSH Terms: conditions — Low Back Pain | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): 1. Give the physical therapy of low back pain educational video + therapist introduction and recommendation video, at the first time of clinic visit.
  2. Physical therapy with hot packing + interference current therapy + pelvic traction + therapeutic exercise, 3 times per week for 4 weeks.
  Interventions: Behavioral: intervention; Other: placebo
- placebo (Placebo Comparator): 1. Give the physical therapy of low back pain educational video, at the first time of clinic visit.
  2. Physical therapy with hot packing + interference current therapy + pelvic traction + therapeutic exercise, 3 times per week for 4 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Behavioral: intervention — intervention with recommendation and therapist introduction
  Arms: intervention
Other: placebo — low back pain education, and physical therapy 3 times per week

SUMMARY:
The trust between patients and medical providers is the cornerstone to obtain success treatment. To boost the trust can increase medical prescription compliance, enhance patient satisfaction, and improve the effectiveness of treatment. Otherwise, mistrust between medical providers and patients will result in ineffective treatment and excessive defensive health care. This situation may cause medical dispute and medical resources wasting problems.

Most of treatment complete in a few times of admissions and interventions. So, how to improve the trust between patients and doctors quickly became a more knotty problem. Several studies found that speech (including listening, showing compassion, and take longer to explain), reputation, clothing, offer a newer therapy were more important than age, title, and sex.

However, past researches were restricted to an unclear causal relationship. That is they can't be determined whether good doctor-patient relationship and better trust conditions create a longer visit time, better satisfaction, and good reputation, or vice versa. They also unable to clarify whether the high degree of trust result in improved treatment effects, or good relationship result from good medical outcomes.

Investigators want to design a randomized control trial by giving patients recommendation and physical therapist introductions to enhance the trust of patients to therapists. And this study may verify whether enhance trust between therapists and patients will lead to changes in treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. First time visit to Taoyuan general hospital rehabilitation ward at 2016/07/01~2017/12/31
2. Diagnosis with L spine spondylosis, L spine Herniated Inter-vertebral Disc, or non-acute low back muscle strain
3. Suitable for physical therapy with ( Hot packing + interference current therapy + pelvic traction + therapeutic exercise )
4. most pain score >2

Exclusion Criteria:

1. poor of follow oral order, or patients who can't understand Chinese, including patients with aphasia or dementia
2. patient who can not received 4 weeks of physical therapy
3. other cause of low back pain which can't treatment with physical therapy, including : (Urinary tract stones, infection, rapid progression disease which need immediately operation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Trust score by The Chinese version of the WFPTS(C-WFPTS) between intervention group and placebo group | The first time data collection for individual 5 mins after the intervention.
Success treatment proportion between intervention group and placebo group 4 weeks after intervention | data collection for individual at the 0 and 4th week after clinical visit
  Success treatment is defined as the most pain score decrease from baseline more than 2 degree.
  ( Pain score change from baseline by Visual Analogue Scale after 4 weeks)

SECONDARY OUTCOMES:
Trust score by The Chinese version of the WFPTS(C-WFPTS) between intervention group and placebo group | The second time and third time data collection after 2 weeks and 4 weeks after first clinical visit
Change of pain score with The Chinese version of the Brief Pain Inventory (BPI-C) between intervention group and placebo group | data collection for individual at the0, 2nd and 4th week after clinical visit
  Pain score change from baseline
Change of the compression force to trigger the tenderness point from baseline | data collection for individual at the 0, 2nd and 4th week after clinical visit
  The compression force was measured by IMADA digital force gauge (kgf) In each data collection point(0 , 2nd and 4th week) , we arrange 3 times test and use the average as the measure value.

CONTACTS AND LOCATIONS:
Overall Officials: Huan-Jui Yeh, Principal Investigator — Department of Physical Medicine and Rehabilitation, Taoyuan General Hospital, Ministry of Health and Welfare, Taiwan
Locations (1):
- Taoyuan general hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No